CLINICAL TRIAL: NCT07032688
Title: A Clinical Study to Evaluate the Pharmacokinetic and Pharmacodynamics Properties of of SHR-3167 Injection at Steady State in Subjects With Type 2 Diabetes
Brief Title: A Clinical Study to Evaluate the Pharmacokinetic and Pharmacodynamics Properties of of SHR-3167 in Subjects With Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-3167-103
Record Dates: First submitted 2025-06-16; First posted 2025-06-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-3167 Group (Experimental)
  Interventions: Drug: SHR-3167 Injection; Drug: Insulin Degludec Injection

INTERVENTIONS:
Drug: SHR-3167 Injection — SHR-3167 injection.
Drug: Insulin Degludec Injection — Insulin Degludec injection.

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics and pharmacodynamics of SHR-3167 at steady state in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities.
2. Age 18~59 years at screening (including cut-off values at both ends).
3. Confirmed diagnosis of type 2 diabetes mellitus ≥ 6 months before screening.
4. Female subjects of childbearing potential and their partners are male subjects of childbearing potential, who have no fertility plan and agree to take high-efficiency contraceptive measures within 3 months after signing the informed consent form and have no plans to donate eggs/sperm; Female subjects of childbearing potential have a negative pregnancy test during the screening period and are not lactating.

Exclusion Criteria:

1. Poor blood pressure control at screening.
2. Known or suspected allergy to investigational drug products or related products; or a history of multiple and/or severe allergies to drugs or foods.
3. Serious cardiovascular and cerebrovascular diseases within 6 months prior to screening.
4. Positive test for hepatitis B surface antigen (HBsAg), HIV antibody, treponema pallidum specific antibody, or hepatitis C virus antibody; or the investigator judges that the subject is in the incubation or active phase of the above infection.
5. Malignancy or history of malignancy within 5 years prior to screening.
6. Participation in any clinical trial of an approved or unapproved investigational drug/medical device within 90 days prior to screening.
7. Any other condition judged by the investigator to be likely to affect the subject's safety or interfere with the evaluation of trial results.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Area under the SHR-3167 concentration-time curve (AUC SHR-3167, tau, ss). | From 0 to 168 hours after SHR-3167 administration.

SECONDARY OUTCOMES:
Maximum observed SHR-3167 concentration (Cmax, ss). | From 0 to 168 hours after SHR-3167 administration.
Adverse events (AEs). | 21 weeks to 43 weeks.
Hypoglycemic events. | 21 weeks to 43 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided